CLINICAL TRIAL: NCT01606982
Title: A Multicenter, Single-arm, Open Label Treatment Protocol to Provide Expanded Access to MDV3100 and Monitor Its Safety in Patients With Progressive Castration-Resistant Prostate Cancer Previously Treated With Docetaxel-Based Chemotherapy
Brief Title: Provide Expanded Access to MDV3100 and Monitor Its Safety in Patients With Progressive Castration-Resistant Prostate Cancer Previously Treated With Docetaxel-Based Chemotherapy
Status: Approved for marketing | Type: Expanded Access
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9785-CL-0401
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: prostate; MDV3100; cancer
MeSH Terms: conditions — Neoplasms | interventions — enzalutamide

INTERVENTIONS:
Drug: MDV3100 — oral
  Other Names: Xtandi; enzalutamide (USAN)

SUMMARY:
The purpose of this treatment protocol is to provide expanded access to MDV3100 and monitor its safety in patients with metastatic castration-resistant prostate cancer previously treated with docetaxel-based chemotherapy.

DETAILED DESCRIPTION:
THE UNITED STATES FOOD AND DRUG ADMINISTRATION (FDA) AND HEALTH CANADA HAVE APPROVED MDV3100 (ENZALUTAMIDE) FOR SALE TO THE PUBLIC, ENROLLMENT IS CLOSED IN BOTH THE UNITED STATES AND CANADA.

The expanded access treatment protocol is being conducted while marketing approval of enzalutamide is being sought. There is no age requirement.

Subjects will complete visits on Day 1, Week 4, Week 12 and then every subsequent 12 weeks until discontinued from the study.

The study will end if enzalutamide is approved for sale to the public by the country's health authority (commercially available) or if the sponsor otherwise decides or is required to end the study. If a subject would like to receive enzalutamide after the study ends, he and the doctor will decide if he should receive a prescription for enzalutamide, with a goal of avoiding any interruption in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) analogue (agonist or antagonist) or orchiectomy
* At least one prior chemotherapy regimen for metastatic castration-resistant prostate cancer with at least one regimen containing docetaxel
* Progressive disease as evidenced by prostate specific antigen (PSA) rise or radiographic or clinical worsening of disease
* No known or suspected brain metastasis
* There is no comparable or satisfactory alternative therapy to treat the subject's disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* History of seizure or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumors, brain metastases, or alcoholism
* History of loss of consciousness or transient ischemic attack within the last 12 months
* Clinically significant cardiovascular disease
* Following lab values:

  * Absolute neutrophil count is <1,000/µL
  * Platelet count is <50,000/µL
  * Hemoglobin is < 5.6 mmol/L (9 g/dL)
  * Total bilirubin ≥1.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≥2.5 x ULN
  * Creatinine clearance is less than 30 ml/min by the Cockcroft and Gault formula
* Subject's conditions suggests that a bone fracture or complication of a bone fracture (such as compression of the spinal cord or other nerves) is likely to occur very soon
* Subject has participated in a previous clinical study of MDV3100 for which the primary endpoint has not yet been reported (e.g., the PREVAIL trial)

Sex: Male
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Derived] Joshua AM, Shore ND, Saad F, Chi KN, Olsson CA, Emmenegger U, Scholz M, Berry W, Mukherjee SD, Winquist E, Haas NB, Foley MA, Dmuchowski C, Perabo F, Hirmand M, Hasabou N, Rathkopf D; Enzalutamide Expanded Access Study Investigators. Safety of enzalutamide in patients with metastatic castration-resistant prostate cancer previously treated with docetaxel: expanded access in North America. Prostate. 2015 Jun;75(8):836-44. doi: 10.1002/pros.22965. Epub 2015 Feb 14. PMID 25683285
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=23